CLINICAL TRIAL: NCT07059754
Title: A Prospective, Feasibility, Single-Center, Clinical Study to Evaluate the Effect of the ETX-4143 Topical Ophthalmic Cooling Device on Ocular Surface Structures and Cell Population in Patients With Chronic Ocular Surface Pain
Brief Title: A Clinical Study to Determine What Effect the EyeCool Treatment Has on the Eye's Surface Anatomy and Inflammation Response After Being Treated for Having Chronic Ocular Surface Pain (COSP)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EyeCool Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETX4143-A005
Record Dates: First submitted 2025-03-29; First posted 2025-07-11 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Eye Pain
Keywords: Chronic Ocular Surface Pain; Ophthalmic Cooling; Topical Ophthalmic Cooling; Cooling Device; Ocular Surface
MeSH Terms: conditions — Eye Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Eyes that are treated with the ETX-4143 topical ophthalmic cooling device
  Interventions: Device: Topical Ophthalmic Cooling

INTERVENTIONS:
Device: Topical Ophthalmic Cooling — Targeted topical ophthalmic cooling treatment using the ETX-4143 cooling device

SUMMARY:
The goal of this clinical trial is to understand what effect a cold treatment with an investigational device, ETX-4143, has on the anatomical structures and the inflammatory response of the surface of the eye in those people who suffer from chronic ocular surface pain (COSP). The trial will also tell us more about the safety of this investigational device. The main questions this study aims to answer are:

* What anatomical changes happen to corneal surface nerves after treatment with ETX-4143
* What changes in inflammatory mediators and cell response take place after treatment with ETX-4143

Researchers will obtain images of the corneal surface nerves for analysis using a confocal microscope and collect tear bio samples for analysis.

Participants will:

* Be screened for having chronic ocular surface pain
* Will be treated with ETX-4143 cold treatment for 4 minutes
* Fill out a weekly questionnaire on eye pain for 12 weeks
* Be seen in the clinic 2 weeks, 6 weeks, and 12 weeks after treatment to have images of the corneal surface taken, and to collect a tear bio sample

DETAILED DESCRIPTION:
EyeCool Therapeutics was founded on the hypothesis that a mild ocular surface cooling treatment, delivered through its proprietary cooling device (ETX-4143), can improve the symptoms of chronic ocular surface pain by transiently inhibiting nerve signaling, and potentially reducing ocular surface inflammation, and potentially restoring normal ocular surface nerve function.

The ETX-4143 Device is a handheld medical device that contains an internal frozen (-20° Centigrade) mixture of purified water and glycerol. The ETX-4143 Device does not contain an active pharmaceutical ingredient. The frozen mixture internally cools two metallic probes that contact the conjunctival surface of the patient; there is no direct contact of the ocular surface with the frozen mixture. Prior to placement of the device on the ocular surface, local anesthesia is administered and a custom speculum used to open and insulate the eyelids, as well as promote correct positioning of the Device. A cornea shield is applied to maintain corneal wetness during the procedure. The Device and accessory (speculum) are provided in disposable, single-use packaging.

In this prospective, single-center, single-center clinical study, 5 adult subjects with chronic ocular surface pain will be identified and treated with the ETX-4143 Device (Cooling Device for topical ophthalmic use). The main goal of the study is to further evaluate the device for changes in ocular surface components using in vivo confocal microscopy, and for safety and efficacy. Improvement in self-reported ocular discomfort and clinical safety measures will be evaluated, along with in vivo confocal microscopy of the cornea before and after treatment.

It is anticipated that the learnings from these observations will be used to design future studies of the ETX-4143 device. In this study, five subjects will receive the investigational product (ETX-4143 Device).

The Medical Monitor will evaluate the clinical safety data as it becomes available and no less than on at least a quarterly basis.

All subjects will be followed for a total of 12 weeks. Subjects will have only the worse eye treated, if both eyes meet the inclusion/exclusion criteria. The worse eye will be determined by the investigator based on subjective reporting from the study subject of chronic ocular surface pain and/or other screening assessments in each eye. Both eyes will be assessed for tear osmolarity and imaged using corneal in vivo confocal microscopy at the University of Melbourne, with the untreated eye representing a control.

ELIGIBILITY:
Inclusion Criteria:

* Documented symptoms of COSP pain for at least 3 months
* A score of ≥5 on the single question COP-Q Eye Pain Severity Module
* Able to obtain sufficient quality corneal in-vivo confocal microscopy images

Exclusion Criteria:

* Less than 50% improvement in VAS Eye Pain score after topical 0.5% proparacaine hydrochloride at screening
* Subjects with clinically significant corneal scarring that could limit the confocal microscopy
* Insufficient number of corneal nerves to permit Fun-IVCM imaging

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Corneal Confocal In-vivo Microscopy Image Analysis | From treatment to the end of twelve weeks
  Non-invasive imaging of the corneal surface for assessing ocular tissue structure.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Casey R VP of Clinical Development, Optometrist, Study Chair — EyeCool Therapeutics, Inc.
Locations (1):
- Sunshine Eye Surgeons, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galor A, Hamrah P, Haque S, Attal N, Labetoulle M. Understanding chronic ocular surface pain: An unmet need for targeted drug therapy. Ocul Surf. 2022 Oct;26:148-156. doi: 10.1016/j.jtos.2022.08.005. Epub 2022 Aug 13. PMID 35970433